CLINICAL TRIAL: NCT06789796
Title: A Randomized, Double-blind Phase III Clinical Study of QL1706 Versus QL1604 as Consolidation Treatment in Patients With Limited-stage Small Cell Lung Cancer Who Have Not Experienced Disease Progression After Concurrent or Sequential Chemoradiotherapy.
Brief Title: a Study of QL1706 or QL1604 in Patients With Limited-stage Small Cell Lung Cancer After Chemoradiotherapy.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1706-310
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 group (Experimental): Iparomlimab and Tuvonralimab + placebo for QL1604, intravenous infusion (IV), every 3 weeks
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706); Drug: placebo for QL1604
- QL1604 group (Active Comparator): QL1604 + placebo for Iparomlimab and Tuvonralimab, IV, every 3 weeks
  Interventions: Drug: QL1604; Drug: placebo for Iparomlimab and Tuvonralimab (QL1706)

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706) — 5mg/kg , every 3 weeks
  Arms: QL1706 group
Drug: placebo for QL1604 — every 3 weeks
  Arms: QL1706 group
Drug: QL1604 — 200mg, every 3 weeks
  Arms: QL1604 group
Drug: placebo for Iparomlimab and Tuvonralimab (QL1706) — every 3 weeks
  Arms: QL1604 group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of QL1706 versus QL1604 monotherapy as consolidation treatment in patients with limited-stage small cell lung cancer (LS-SCLC) who have not experienced disease progression after concurrent or sequential chemoradiotherapy.

QL1706 (Iparomlimab and Tuvonralimab) is a single bifunctional MabPair product against PD-1 and CTLA-4. QL1604 is a monoclonal antibody against PD-1.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be aged between 18 and 75 years (inclusive of boundary values), and both males and females are eligible.
* Pathologically confirmed LS-SCLC [I-III stage SCLC (any T, any N, M0)], according to the American Joint Committee on Cancer (AJCC, 8th edition) staging manual.
* Received 4 cycles of chemotherapy concurrent or sequential with radiotherapy. Chemotherapy must contain platinum and etoposide. Radiotherapy must be either total 60-70 Gy over 6 weeks for the QD regimen or total 45 Gy over 3 weeks for BID schedules.
* Patients must have achieved a complete response (CR), partial response (PR), or stable disease (SD) after receiving curative platinum-based CRT and must not have developed progressive disease (PD) prior to study entry.

Exclusion Criteria:

* Mixed SCLC and non-small cell lung cancer (NSCLC).
* Extensive-stage SCLC.
* Active or prior documented autoimmune or inflammatory disorders.
* Received other chemotherapy regimens besides etoposide and platinum-based therapy.
* Active or prior documented autoimmune or inflammatory disorders.
* Presence of interstitial lung disease or active non-infectious pneumonia (excluding grade 1 radiation pneumonitis not treated with corticosteroids).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after chemoradiotherapy (CRT) for patients with LS-SCLC as measured by Blinded Independent Review Committee (BIRC)-assessed PFS
Overall survival (OS) | up to 5 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by OS

SECONDARY OUTCOMES:
objective response rate (ORR) | up to 2 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by ORR
disease control rate (DCR) | up to 2 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by DCR
duration of response (DoR) | up to 2 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by DoR
PFS | up to 2 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by Investigator-assessed PFS
1-year OS rate | up to 1 year
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by 1-year OS rate
2-year OS rate | up to 2 years
  To compare and evaluate the efficacy of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by 2-year OS rate
adverse events | up to 2 years
  To compare and evaluate the safety of QL1706 versus QL1604 as consolidation therapy after CRT for patients with LS-SCLC as measured by the incidence of adverse events (Percentage of participants with treatment-related adverse events as assessed by CTCAEv5.0.) and abnormal laboratory parameters.